CLINICAL TRIAL: NCT05749042
Title: Concurrent Chemoradiotherapy Based of Cisplatin With or Without Sintilimab as First-line Therapy for Patients With Advanced Oral Cavity Squamous Cell Carcinoma :a Phase 2,Prospective, Open-label,Unicentral,Randomised Controlled Trial
Brief Title: A Study of Concurrent Chemoradiotherapy Based of Cisplatin With or Without Sintilimab as First-line Therapy for Patients With Advanced Oral Cavity Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTGU006
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — sintilimab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab+Cisplatin+Radiotherapy (Experimental)
  Interventions: Drug: Sintilimab
- Cisplatin+Radiotherapy (Active Comparator)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Concurrent Chemoradiotherapy Based of Cisplatin Plus Sintilimab.
  Other Names: Cisplatin; Radiotherapy
  Arms: Sintilimab+Cisplatin+Radiotherapy
Radiation: Radiotherapy — Concurrent Chemoradiotherapy Based of Cisplatin
  Other Names: Cisplatin
  Arms: Cisplatin+Radiotherapy

SUMMARY:
This study aims to evaluate the efficacy and safety of concurrent chemoradiotherapy based of cisplatin with sintilimab as first-line therapy for patients with advanced oral cavity squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign informed consent.
2. Age ≥18 years, and ≤75years , either sex.
3. Eastern Collaborative Oncology Group Performance status (ECOG PS) 0 ,1 or 2.
4. Eastern Collaborative Oncology Group Performance status (ECOG PS) 0 ,1 or 2.
5. Patients with oral squamous cell carcinoma (including gingival cancer, tongue cancer, lip cancer, buccal cancer, oral cancer, etc) diagnosed by histopathology (according to the 8th edition of AJCC).
6. Initial diagnosis patients unable to perform surgery.
7. Have at least one measurable lesion as defined by RECIST 1.1.
8. Normal hepatic function: total bilirubin≤1.5×normal upper limit (ULN); Alanine aminotransferase and Aspartate aminotransferase levels ≤2.5×ULN or ≤5×ULN if liver metastasis is present.
9. Normal renal function ：Creatinine ≤1.5×ULN or calculated creatinine clearance ≥45 mL/min (using Cockcroft/Gault formula to calculate ).
10. Normal hematological function：absolute neutrophil count ≥1.5×109/L, platelet count ≥70×109/L, hemoglobin≥80g/L [no blood transfusion or erythropoietin (EPO) within 7 days] Dependency].
11. Has a life expectancy of at ≥3 months.

Exclusion Criteria:

1. ECOG PS >2.
2. Patients who received radiotherapy, chemotherapy, monoclonal antibody and oral EGFR-TKI therapy within three months.
3. Patients who are receiving any other investigational agents within 30 days prior to entering the study.
4. The tumor has metastasized to the brain and / or pia mater.
5. History of other malignancies (except for cured cervical carcinoma in situ or skin basal cell carcinoma and other malignancies that have been cured for more than 5 years).
6. Accompanied by other serious diseases, including but not limited to:

   Uncontrollable congestive heart failure (NYHA grade Ⅲ or Ⅳ), unstable angina, poorly controlled arrhythmia, uncontrolled moderate or above hypertension (SBP > 160mmhg or DBP > 100mmhg) ; Severe active infection; Uncontrollable diabetes (refers to the high fluctuation of blood glucose, the impact on patients' life and the frequent occurrence of hypotension despite the standard insulin treatment and frequent blood glucose monitoring) ; Mental illness affecting informed consent and / or program compliance.
7. Those who are allergic to the drug or its components used in the program.
8. Pregnancy (confirmed by hCG test in blood or urine) or lactating women, or childbearing age subjects are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last trial treatment.
9. Those who are not considered suitable for the study by the researchers.
10. Unwilling to participate in this study or unable to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Compare Progression Free Survival (PFS) between Chemoradiotherapy Based of Cisplatin + Sintilimab Regimen and Chemoradiotherapy Based of Cisplatin Regimen using RECIST 1.1. | approximately 24 months
  PFS was defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1.
Compare objective response rate(ORR) between Chemoradiotherapy Based of Cisplatin + Sintilimab Regimen and Chemoradiotherapy Based of Cisplatin Regimen using RECIST 1.1. | approximately 24 months
  ORR was defined as the percentage of participants with confirmed objective tumor response, complete response (CR) or partial response (PR), as determined by investigator using RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Compare Overall Survival (OS) between Chemoradiotherapy Based of Cisplatin + Sintilimab Regimen and Chemoradiotherapy Based of Cisplatin Regimen. | approximately 24 months
  Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. Data for participants who were not reported as dead at the time of analysis was censored at the date when they were last known to be alive.
Compare Disease Control Rate (DCR) between Chemoradiotherapy Based of Cisplatin + Sintilimab Regimen and Chemoradiotherapy Based of Cisplatin Regimen using RECIST 1.1. | approximately 24 months
  DCR was defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, Hubei, China

IPD SHARING:
Plan to Share IPD: No